CLINICAL TRIAL: NCT06155396
Title: A Single-Arm, Open- Label, Multicenter Phase II Study of RC48-ADC in Combination With Zimberelimab Injection for the Treatment ,at Least First-line Platinum-containing Standard Therapy Failed in HER2-expressing Subject With Recurrent or Metastatic Cervical Cancer
Brief Title: A Study of RC48-ADC Combination With Zimberelimab Injection Therapies at Least First-line Platinum-containing Standard Therapy Failed With Recurrent or Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C030
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer
Keywords: HER2-expressing; Recurrent Cervical Cancer; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — disitamab vedotin; zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin + Zimberelimab (Experimental): Disitamab Vedotin（RC48-ADC）with Zimberelimab arm
  Interventions: Drug: Disitamab Vedotin; Drug: Zimberelimab

INTERVENTIONS:
Drug: Disitamab Vedotin — 2.0 mg/kg IV every 2 weeks
  Other Names: Disitamab Vedotin （RC48-ADC)
Drug: Zimberelimab — 240mg IV every 2 weeks

SUMMARY:
This study will evaluate the efficacy,safety of RC48-ADC in Combination with Zimberelimab Injection for the Treatment ,at least first-line platinum-containing standard therapy failed in HER2-expressing subject with Recurrent or Metastatic Cervical Cancer

DETAILED DESCRIPTION:
This is a Phase II, Single-Arm ,multicenter, open-label clinical trial designed to evaluate safety and efficacy of RC48-ADC in Combination with Zimberelimab Injection for the Treatment ,at least first-line platinum-containing standard therapy failed in HER2-expressing subject with Recurrent or Metastatic Cervical Cancer.The HER2-expressing is defined as: the HER2 IHC 3+ or 2+, or 1+.subjects with IHC 2+ require testing for FISH.

ELIGIBILITY:
Inclusion Criteria:

1. a)Patients with histologically confirmed HER2-expressing recurrent or metastatic cervical cancer who have failed at least 1 line of standard platinum-containing therapy ; b) Not suitable for surgery or radiotherapy;
2. Voluntarily agreed to participate in the study and signed an informed consent form.
3. Female, age ≥ 18 years
4. Expected survival ≥ 12 weeks
5. Central laboratory confirmation of HER2 expression: IHC 1+, 2+, or 3+; subjects with IHC 2+ require testing for FISH.
6. Central laboratory confirmation of PD-L1 expression
7. Measurable disease according to RECIST 1.1 standard
8. ECOG physical condition 0 or 1 point
9. Adequate organ function, criteria should be met during the screening period

   1. ANC ≥1,500/µL
   2. platelet count ≥100,000/μL
   3. hemoglobin ≥9.0 g/dL
   4. total bilirubin ≤1.5 × upper limit normal (ULN) OR direct bilirubin ≤ULN for subjects with total bilirubin >1.5 × ULN. Serum bilirubin ≤3× ULN for subjects with Gilbert's disease
   5. CrCl ≥50 mL/min (measured by the Cockcroft-Gault formula as applicable, or 24-hour urine).
   6. ALT and AST ≤2.5× ULN without liver metastases or ≤5× ULN with liver metastases
   7. LVEF ≥>50%
10. Female subjects should be surgically sterilised, post-menopausal or agree to use at least one medically approved contraceptive method during and for 6 months after the end of the study treatment period, must have had a negative blood pregnancy test within 7 days prior to study entry, and must be non-lactating.
11. Willingness and ability to comply with trial and follow-up procedure arrangements.

Exclusion Criteria:

1. Have central nervous system metastases and/or carcinomatous meningitis.
2. Received anti-tumour therapy or participated in another clinical study treatment within 4 weeks prior to the start of study treatment.
3. Toxicity due to previous antineoplastic therapy has not recovered to NCI-CTCAE (version 5.0) grade 0-1.
4. Major surgery with incomplete recovery within 4 weeks prior to start of study dosing.
5. Serum virology examination (based on the normal value of the research center) :

   1. HBsAg test results were positive, and HBV DNA copy number was positive;
   2. HCVAb test results were positive (HCV RNA PCR test results were negative only to be included in this study);
   3. HIVAb tested positive
6. Have received a live or live attenuated vaccine within 4 weeks prior to the start of study dosing; or plan to receive any vaccine during the study period
7. Grade 3 or higher heart failure
8. History of gastrointestinal perforation and/or fistula within the previous 6 months
9. Serious arterial/venous thrombotic event or cardiovascular accident within 1 year prior to study drug administration
10. Presence of active or progressive infection requiring systemic therapy, with severe infection within 4 weeks prior to first dose;
11. Active TB.
12. Presence of systemic disease not under stable control as judged by the investigator.
13. History of interstitial pneumonia, obstructive lung disease, drug-induced pneumonia, radiation pneumonia, idiopathic pneumonia or active pneumonia.
14. Clinically relevant pyelonephrosis cannot be alleviated by ureteral stents or percutaneous drainage.
15. Presence of active autoimmune disease requiring systemic therapy within 2 years prior to the start of study drug administration, allowing for relevant alternative therapy.
16. Other malignancy within 5 years prior to start of study drug administration.
17. Previous allogeneic haematopoietic stem cell transplantation.
18. Previous treatment with other Antibody-drug conjugateantibody-coupled drugs.
19. Known hypersensitivity to the drug vedicilizumab for injection and its components or to Zimberelimab injection and other monoclonal antibodies.
20. Have any other disease, metabolic abnormality, physical examination abnormality or laboratory test abnormality.
21. Estimated lack of patient adherence to participate in this clinical study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety run-in ：Safety(adverse event) | Up to approximately 2 years
  to evaluate safety including adverse event rate and adverse event grade.
Dose extension period ：Objective Response Rate (ORR) | Up to approximately 2 years
  The objective response rate will be mainly analyzed by according to the RECIST 1.1 standard tumor evaluation by the investigator will be performed

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | Up to approximately 2 years
  The objective response rate will be mainly analyzed by according to the RECIST 1.1 standard tumor evaluation by the investigator will be performed
Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease Control Rate(DCR) | Up to approximately 2 years
  Proportion of patients whose tumors shrank or stabilized for a certain period of time
Progression-free survival (PFS), evaluated by the investigator | Up to approximately 2 years
  Progression-free survival (PFS) refers to the time from the date of first administration to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.
Overall survival (OS) | Up to approximately 2 years
  Overall survival (OS) refers to the time from the date of first administration to the date of death of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (12):
- China (12):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Beijing Obstetrics and Gynecology Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangxi Tumor Hospital, Nanning, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No